CLINICAL TRIAL: NCT02231606
Title: Potentiating Rural Investment in Children's Eyecare (PRICE)
Acronym: PRICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Orbis (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); The Fred Hollows Foundation (Unknown); Rural Education Action Project (Unknown); Second People's Hospital of Yunnan Province (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Professor, MD,MPH, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ZOC-PRICE
Record Dates: First submitted 2014-08-31; First posted 2014-09-04 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Myopia
Keywords: Myopia Prevalence; Proportion of Purchase of free Spectacles; Proportion of Purchase of update Spectacles; Proportion of Wearing Spectacles
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Pure Control (No Intervention): Provision of glasses prescription only
- Group 2: Free Glasses (Experimental): Free glasses for all, no upgrade glasses offered
  Interventions: Other: Free Glasses
- Group 3: Free + Upgrade Glasses 1 (Experimental): Free glasses for all, optional purchase from range of spectacles, cheapest RMB100 (Mean price paid for glasses by Control families in Seeing is Learning I, subtracting one SD)
  Interventions: Other: Free Glasses; Other: Upgrade Glasses 1
- Group 4: Free + Upgrade Glasses 2 (Experimental): Free glasses for all, optional purchase from range of spectacles, cheapest RMB200 (Mean price paid for glasses by Control families in Seeing is Learning I, adding one SD)
  Interventions: Other: Free Glasses; Other: Upgrade Glasses 2

INTERVENTIONS:
Other: Free Glasses — Provide free glasses
  Arms: Group 2: Free Glasses; Group 3: Free + Upgrade Glasses 1; Group 4: Free + Upgrade Glasses 2
Other: Upgrade Glasses 1 — Provide optional purchase from range of spectacles, cheapest RMB100 (Mean price paid for glasses by Control families in Seeing is Learning I, subtracting one SD)
  Arms: Group 3: Free + Upgrade Glasses 1
Other: Upgrade Glasses 2 — Provide optional purchase from range of spectacles, cheapest RMB200 (Mean price paid for glasses by Control families in Seeing is Learning I, adding one SD)
  Arms: Group 4: Free + Upgrade Glasses 2

SUMMARY:
The aim of the project is to create, study and advocate for a model that can be adopted by the Chinese government to provide spectacles for all children sustainable.

DETAILED DESCRIPTION:
Uncorrected refractive error (URE) is the leading cause of visual impairment among Chinese children, accounting for 90% or more of poor vision, and Chinese children have among the highest rates of myopia in the world. Despite the fact that the problem of URE is safely and inexpensively treated with glasses, only 15-40% of children needing them own and wear glasses sufficient to provide good vision in rural China.

PRICE (Potentiating Rural Investment in Children's Eyecare) will use a randomized, controlled design across 4 groups of all 138 schools in Yunnan (one of China's poorest provinces) and Guangdong (one of the richest) to optimize the model of "free glasses for all with an optional upgrade." The selection of free spectacles and cost of the "upgrade" options will be varied between groups in order to find the optimal balance between high rates of purchase of upgrade glasses on the one hand and good acceptance and wear of free spectacles among those selecting them on the other.

ELIGIBILITY:
Inclusion Criteria:

1. Randomly selected primary schools, which has all 3, 4 and 5 grades, in the 9 project counties.
2. A class randomly selected from each grade of 3, 4, and 5 grades of the selected primary schools.
3. All children in the selected classes.

Exclusion Criteria:

1. Those schools that the total number of students are more than 2000.
2. Those schools that the total number of students of 3, 4, 5 grades are less than 80.
3. Children suffering from eye diseases such as cataract, congenital ptosis, strabismus, congenital glaucoma will not be included in the study and will be recommended referral.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10234 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Glasses purchase proportion | 8 months after the start of the project.
  Proportion of children in each group requiring glasses whose families select to purchase them.

SECONDARY OUTCOMES:
Wearing spectacles proportion | 8 months after the start of the project.
  Proportion of children who actually wearing glasses at an unannounced check at endline survey.

OTHER OUTCOMES:
Visual acuity | At the first week of the study, two months later, and six months later.
  There are three times of vision acuity(VA) check. The baseline VA, the fraction VA and the endline VA with and without glasses
Mydriatic refraction results | One month after visual screening.
  Those uncorrected VA ≤ 6/12 in either eye and 25% of the students whose uncorrected VA > 6/12 in both eyes will receive mydriatic refraction.
Family economic conditions | At the first week of the study
  Collect the children's family economic information on baseline survey.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — The Key Laboratory, Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] He M, Zeng J, Liu Y, Xu J, Pokharel GP, Ellwein LB. Refractive error and visual impairment in urban children in southern china. Invest Ophthalmol Vis Sci. 2004 Mar;45(3):793-9. doi: 10.1167/iovs.03-1051. PMID 14985292
- [Background] Zhou Z, Zeng J, Ma X, Pang X, Yi H, Chen Q, Meltzer ME, He M, Rozelle S, Congdon N. Accuracy of rural refractionists in western China. Invest Ophthalmol Vis Sci. 2014 Jan 7;55(1):154-61. doi: 10.1167/iovs.13-13250. PMID 24327616
- [Background] Li L, Lam J, Lu Y, Ye Y, Lam DS, Gao Y, Sharma A, Zhang M, Griffiths S, Congdon N. Attitudes of students, parents, and teachers toward glasses use in rural China. Arch Ophthalmol. 2010 Jun;128(6):759-65. doi: 10.1001/archophthalmol.2010.73. PMID 20547954
- [Background] He M, Zheng Y, Xiang F. Prevalence of myopia in urban and rural children in mainland China. Optom Vis Sci. 2009 Jan;86(1):40-4. doi: 10.1097/OPX.0b013e3181940719. PMID 19104465
- [Derived] Wang X, Congdon N, Ma Y, Hu M, Zhou Y, Liao W, Jin L, Xiao B, Wu X, Ni M, Yi H, Huang Y, Varga B, Zhang H, Cun Y, Li X, Yang L, Liang C, Huang W, Rozelle S, Ma X. Cluster-randomized controlled trial of the effects of free glasses on purchase of children's glasses in China: The PRICE (Potentiating Rural Investment in Children's Eyecare) study. PLoS One. 2017 Nov 21;12(11):e0187808. doi: 10.1371/journal.pone.0187808. eCollection 2017. PMID 29161286